CLINICAL TRIAL: NCT06978231
Title: Effect of Same-session Endoscopic Ultrasonography on Endoscopic Retrograde Cholangiopancreatography in Pancreaticobiliary Diseases: A Randomized Controlled Trial
Brief Title: Effect of Same-session EUS on ERCP in Pancreaticobiliary Diseases
Acronym: EUS、 ERCP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025SDU-QILU-3
Record Dates: First submitted 2025-05-10; First posted 2025-05-18 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-06

CONDITIONS: Pancreaticobiilary Diseases
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EUS+ERCP group (Experimental): EUS and ERCP were performed during the same session under continuous sedation/anesthesia in the intervention group.
  Interventions: Procedure: EUS+ERCP
- ERCP group (Other): Only ERCP was performed in the control group
  Interventions: Procedure: ERCP

INTERVENTIONS:
Procedure: EUS+ERCP — EUS were performed during the same session with ERCP under continuous sedation/anesthesia
  Arms: EUS+ERCP group
Procedure: ERCP — Only ERCP was performed in the control group
  Arms: ERCP group

SUMMARY:
This is a single-center randomized controlled trial. Eligible subjects meeting inclusion/exclusion criteria will be randomized 1:1 to EUS+ERCP group or ERCP group. Clinical data and patient-reported outcomes are regularly collected at baseline and during follow-up periods. A comparative analysis was conducted to assess the impact of same-session EUS on ERCP strategy modification between two groups, utilizing a structured questionnaire.Secondarily, the safety and efficacy of same-session EUS will be comprehensively evaluated by comparing complication rates, technical success rate and hospitalization costs, length of stay, and radiation exposure between groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years;
2. Patients with pancreaticobiliary diseases definitively indicated for ERCP (as confirmed by HBP Specialists );
3. No prior history of ERCP;
4. No pancreaticobiliary EUS examinations within the preceding 3 months.

Exclusion Criteria:

1. Patients with clinically confirmed malignant lesions deemed surgically unresectable by multidisciplinary evaluation and requiring pathological diagnosis exclusively for chemotherapy/radiotherapy guidance;
2. Patients with confirmed diagnosis requiring only palliative biliary/pancreatic stent placement for obstructive jaundice ;
3. Patients with anatomical alterations or surgical history affecting EUS feasibility;
4. Severe systemic illness including severe hepatic, renal, cardiopulmonary and cerebrovascular diseases with high risk for endoscopic procedures;
5. Contraindication to iodinated contrast media (allergy or renal impairment preventing ERCP);
6. Pregnancy or lactation;
7. Patients with severe coagulopathy;
8. Declined informed consent;
9. Severe psychiatric disorder/non-cooperation precluding safe procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
ERCP strategy modification rate | From enrollment to 6 months after the end of treatment
  Concordance rate between anticipated and actual ERCP procedural strategies and the rate of avoiding unnecessary ERCP procedures.

SECONDARY OUTCOMES:
Procedure outcomes | From enrollment to 6 months after the end of treatment
  Technical success rate (defined as successful completion of intended therapeutic intervention) ERCP procedure time (from duodenoscope insertion to withdrawal) Difficult cannulation rate (requiring advanced techniques or >5 attempts)
Incidence of complications | From enrollment to 6 months after the end of treatment
Radiation-related situation | From enrollment to 6 months after the end of treatment
  Fluoroscopy time (minutes) Radiation exposure (dose-area product, Gy·cm²)
Healthcare utilization measures | From enrollment to 6 months after the end of treatment
  Hospital length of stay (days) Total hospitalization costs

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No